CLINICAL TRIAL: NCT01442090
Title: A Phase II, Open-Label, Randomized Study of GDC-0980 Versus Everolimus in Patients With Metastatic Renal Cell Carcinoma Who Have Progressed on or Following VEGF-Targeted Therapy
Brief Title: Study of GDC-0980 Versus Everolimus in Participants With Metastatic Renal Cell Carcinoma Who Have Progressed on or Following Vascular Endothelial Growth Factor- (VEGF) Targeted Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIM4973g; GO00885 (Other: Hoffmann-La Roche); 2011-000493-56 (EudraCT Number)
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-05

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus; 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one

ARMS (2):
- Everolimus (Active Comparator): Participants will receive everolimus (10 mg) orally daily until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: Everolimus
- GDC-0980 (Experimental): Participants will receive GDC-0980 (40 mg) orally daily until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: GDC-0980

INTERVENTIONS:
Drug: Everolimus — Everolimus will be administered orally at a 10 mg daily dose.
  Arms: Everolimus
Drug: GDC-0980 — GDC-0980 will be administered orally at a 40 mg daily dose.
  Arms: GDC-0980

SUMMARY:
Study PIM4973g is a multicenter, international, open-label Phase II trial. Participants with metastatic renal cell carcinoma who have progressed on or after VEGF targeted therapy will be randomized in 1:1 to two groups either to receive daily GDC-0980 or everolimus orally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable metastatic renal cell carcinoma with clear-cell component that progressed on or within 6 months of stopping VEGF-targeted therapy
* Disease that is measurable per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
* Karnofsky performance status of greater than or equal to (>=) 70 percent (%)
* Adequate hematologic and end organ function
* For female participants of childbearing potential and male participants with partners of childbearing potential, agreement to use two effective forms of contraception and to continue its use for the duration of the study

Exclusion Criteria:

* Any anti-cancer therapy, including chemotherapy, biologic or other targeted therapy, herbal therapy, hormonal therapy, or radiotherapy, within 5 half-lives (for systemic agents) or 2 weeks, whichever is shorter, prior to Day 1. Certain forms of radiation therapy may be considered for pain palliation if participants are deriving benefit
* Previously established diagnosis of pulmonary fibrosis of any cause
* New York Heart Association (NYHA) Class II or greater congestive heart failure
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Presence of positive test results for hepatitis B (hepatitis B [HB] surface antigen [HBsAg] and/or total HB core antibody [anti-HB-c; both tests are required]) or hepatitis C
* Known human immunodeficiency virus (HIV) infection
* Pregnancy, lactation, or breastfeeding
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment
* Leptomeningeal disease as a manifestation of cancer
* History of other malignancies less than equal to <= 5 years of Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Need for current chronic corticosteroid therapy (>= 10 milligrams [mg] of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids for greater than [>] 7 days) or use of other immunosuppressant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
DUration of progression-free survival (PFS) as assessed by the investigator using RECIST v1.1 | Baseline until disease progression or death, whichever occurred first (up to approximately 23 months)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of GDC-0980 | pre-dose and 1, 2, 4 hours post-dose on Week 1 Day 1, Pre-dose on Week 1 Day 2, pre-dose and 2 hours post dose on Week 3 Day 1 and Week 9 Day 1, 48 hours after last dose (up to approximately 23 months)
Cmax of everolimus | pre-dose and 2, hours post-dose on Week 1 Day 1 and Week 9 Day 1, 48 hours after last dose (up to approximately 23 months)\n
Minimum plasma concentration (Cmin) of GDC-0980 | pre-dose on Week 1 Day 1, Week 1 Day 2, Week 3 Day 1 and Week 9 Day 1
Cmin of everolimus | pre-dose on Week 1 Day 1 and Week 9 Day 1
Number of participants with adverse events | up to 30 days after end of treatment (approximately up to 23 months)
Number of participants with objective tumor response as assessed by the investigator using RECIST v1.1 | Baseline until disease progression or death, whichever occurred first (up to approximately 23 months)
Duration of objective tumour response as assessed by the investigator using RECIST v1.1 | Baseline until disease progression or death, whichever occurred first (up to approximately 23 months)
Duration of overall survival (OS) | Baseline until death (up to approximately 45 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (20):
- United States (8):
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Boston, Massachusetts
  - Las Vegas, Nevada
  - New York, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Nashville, Tennessee
- France (3):
  - Bordeaux
  - Paris
  - Villejuif
- Germany (3):
  - Berlin
  - Hanover
  - München
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid
- United Kingdom (4):
  - Leeds
  - London
  - Manchester
  - Sutton

REFERENCES:
- [Derived] Powles T, Lackner MR, Oudard S, Escudier B, Ralph C, Brown JE, Hawkins RE, Castellano D, Rini BI, Staehler MD, Ravaud A, Lin W, O'Keeffe B, Wang Y, Lu S, Spoerke JM, Huw LY, Byrtek M, Zhu R, Ware JA, Motzer RJ. Randomized Open-Label Phase II Trial of Apitolisib (GDC-0980), a Novel Inhibitor of the PI3K/Mammalian Target of Rapamycin Pathway, Versus Everolimus in Patients With Metastatic Renal Cell Carcinoma. J Clin Oncol. 2016 May 10;34(14):1660-8. doi: 10.1200/JCO.2015.64.8808. Epub 2016 Mar 7. PMID 26951309